CLINICAL TRIAL: NCT01880905
Title: The Length of Uteroovarian Ligament and the Risk of Ovarian Torsion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Amir Wiser, MD, Meir Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0031-13-MMC
Record Dates: First submitted 2013-06-11; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-04

CONDITIONS: Ovarian Torsion
Keywords: the length of uterine ovarian ligament
MeSH Terms: conditions — Ovarian Torsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- female undergoing gynecological surgery (Experimental)
  Interventions: Procedure: Measure of uteroovarian ligament length during gynecological surgery

INTERVENTIONS:
Procedure: Measure of uteroovarian ligament length during gynecological surgery

SUMMARY:
Ovarian torsion is one of the gynecological emergency. This complication requires high clinical suspicion and early detection, to prevent permanent loss of ovarian function. The long uterine ovarian ligament could be a risk factor for ovarian torsion. We want to measure the uterine ovarian ligament length during routine laparoscopy/laparotomy and to compare the length between the torsion group and other non torsion patients

DETAILED DESCRIPTION:
Female patient who are going to undergo laparoscopy/laparotomy for any gynecological reason will ask to participate. During the operation the uteroovarian ligament length will be measure by sterile ruler (calibrated plastic device 1 mm in diameter).

The length of uteroovarian ligament will compared between the patient who will diagnose with ovarian torsion (study group) and the other women (control group)

ELIGIBILITY:
Inclusion Criteria:

* Indication for gynecological operation
* hemodynamically stable

Exclusion Criteria:

* Ovarian torsion in the past
* History of pelvic inflammatory disease (PID)

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
uteroovarian ligament length | 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel